CLINICAL TRIAL: NCT03310827
Title: An Investigation of DNA-based Dietary Advice and Its Effects on Changing Health Behaviours in Adults With Depressive Disorders: A Mixed Methods Study to Evaluate Efficacy and Participant Experiences
Brief Title: DNA-based Dietary Advice for Adults With Depressive Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karen Davison (Other)
Responsible Party: Sponsor-Investigator, Karen Davison, Principal Investigator, Kwantlen Polytechnic University
Organization: Kwantlen Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KK17-01
Record Dates: First submitted 2017-09-20; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: Nutrition; Nutrigenomics
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: a phase I randomized controlled trial of 42 adults (19 to 50 years) with depressive disorders using a 2:1 ratio of group selection (28 in the intervention {I} group and 14 in the control {C} group) is proposed.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Nutrition (Experimental): Participant receives gene test results with diet plan (personalized nutrition)
  Interventions: Behavioral: Personalized Nutrition
- Gene Test Report Only (Placebo Comparator): Participant receives standard diet plan
  Interventions: Behavioral: Personalized Nutrition

INTERVENTIONS:
Behavioral: Personalized Nutrition — Diet plan based on nutrition-related gene test results

SUMMARY:
To evaluate the feasibility of nutrigenomics as an intervention for mental health conditions, a phase I randomized controlled trial of 42 adults (19 to 50 years) with depressive disorders using a 2:1 ratio of group selection (28 in the intervention {I} group and 14 in the control {C} group) is proposed. Participants with a confirmed depressive disorder will be recruited from two local mental health clinics. Those randomized into the I group will do the gene testing and be provided personalized DNA-based dietary advice from a registered dietitian; those in the C group will also receive testing but be given general dietary advice by a registered dietitian. Pre- and post-intervention comparisons (3 and 6 weeks after a personalized nutrition plan is given) will be analyzed based on records of dietary intakes (i.e., 3 day food records and food frequency questionnaire) and psychiatric functioning (e.g., Quick Inventory of Depressive Symptomology, Hospital Anxiety and Depression Scale, Outcome Questionnaire - OQ-45). In addition, measures that track physical activity, sedentary behavior, and sleep quality as well as sociodemographics will be included as covariates. After the intervention study is completed, in-depth focus group interviews will be conducted. Participants will be asked questions that will elicit their perceptions of the nutrigenomics test and the personalized dietary advice provided as well as the behavioural response to disclosure of genetic information.

DETAILED DESCRIPTION:
While evidence suggests that the disclosure of personal genetic information based on nutrigenomics testing leads to lifestyle behaviour changes in selected populations, the potential for its use as an intervention in clinical populations, such as those with depressive disorders, has yet to be explored.

Study Objectives: The proposed study will employ a mixed-methods approach and focus on the following objectives:

1. to examine the efficacy of testing for 12-genes (i.e., CYP1A2, UCP1, MTHFR, HLA, TMPRSS6, TFR2, TF, MCM6, NOS3, ACE, FUT2, GSTT1, TCF7L2) that assess 11 dietary components (i.e, caffeine, energy balance, folate gluten, iron, lactose, omega-3 fat, sodium, vitamin B12, vitamin C, and whole grains) in changing diet quality, eating behaviours and improving symptoms in adults with depressive disorders
2. to conduct a qualitative investigation of participants' experiences with using gene testing that assesses for dietary components

Summary of Method: To evaluate the feasibility of nutrigenomics as an intervention for mental health conditions, a phase I randomized controlled trial of 24 adults with depressive disorders using a 2:1 ratio of group selection (16 in the intervention {I} group and 8 in the control {C} group) is proposed. Participants with a confirmed depressive disorder will be recruited from two local mental health clinics. Those randomized into the I group will do the gene testing and be provided personalized DNA-based dietary advice from a registered dietitian; those in the C group will also receive testing but be given general dietary advice by a registered dietitian. Pre- and post-intervention comparisons (3 and 6 weeks after a personalized nutrition plan is given) will be analyzed based on records of dietary intakes (i.e., 3 day food records and food frequency questionnaire) and psychiatric functioning (e.g., Quick Inventory of Depressive Symptomology, Hospital Anxiety and Depression Scale, Outcome Questionnaire - OQ-45). In addition, measures that track physical activity, sedentary behavior, and sleep quality as well as sociodemographics will be included as covariates.

After the intervention study is completed, in-depth focus group interviews will be conducted. Participants will be asked questions that will elicit their perceptions of the nutrigenomics test and the personalized dietary advice provided as well as the behavioural response to disclosure of genetic information.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are living in the community and 19 years of age or older.
2. Mild to moderate depression as measured by the Quick Inventory of Depressive Symptomology (QIDS10).
3. A level of understanding sufficient to perform all tests and examinations required by the protocol.

Exclusion Criteria:

1. Investigators and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
2. Current or lifetime diagnosis of any of the following according to DSM-IV or DSM-5 criteria: Schizophrenia Spectrum and Other Psychotic Disorders, Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder, Delusional Disorder, Psychotic Disorder Not Otherwise Specified, Delirium of any type, Dementia of any type, Amnestic Disorder, any Substance-Induced Disorder, or any Psychotic Disorder due to a General Medical Condition.
3. Alcohol or drug dependence during the previous 12 months. Participants must have consumed less than 10 alcoholic beverages per week in the previous 4 weeks and had no use of marijuana and other illicit drugs. At each visit, participants will be asked for an estimate of their use of each of these substances, and these amounts will be recorded for possible later statistical analysis.
4. Hospitalization for treatment of a mental health condition within the previous 6 months.
5. Serious, unstable illnesses such that death is anticipated within 1 year or intensive care unit hospitalization for the disease is anticipated within 6 months. This includes hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic diseases (specifically current agranulocytosis with an absolute neutrophil count <500 mm3).
6. Indication of treatment resistance (e.g., has been given more than 3 treatments for depression).
7. Not taking any atypical antipsychotics or anti-depressants that have an appetite stimulating effect (e.g., Mirtazapine)
8. Uncorrected hypothyroidism or hyperthyroidism in the previous 12 months.
9. Diagnosed Inflammatory Bowel Syndrome, or any other chronic gastrointestinal problem.
10. Treatment with electroconvulsive therapy (ECT) within previous 6 months.
11. Patients will be excluded temporarily if they have taken an oral antibiotic in the previous 6 weeks. If an antibiotic is begun during the course of the trial, that patient will be withdrawn from the study.
12. Taking any type of nutritional or herbal supplement, including melatonin, known to have a centrally-acting effect. However, participants who have been taking supplements such as Echinacea, chondroitin, or glucosamine may enter the study if a) they have been taking these agents for at least one month prior to the study, and b) they continue on these agents throughout the study. Supplement information will be presented at intake, and the cessation of any such supplements will be required for the participant to continue in screening.
13. Women who are pregnant or breast-feeding; women of childbearing potential who are not using a medically accepted means of contraception when engaging in sexual intercourse (for example, intrauterine device, oral contraceptive, implant, Depo-Provera, or barrier devices with spermicide). Women who become pregnant during the trial will be withdrawn.
14. Any person judged clinically to be at serious risk for suicide or violence.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Outcome Questionnaire-45 | 3 months
  Measures symptom distress (depression and anxiety), interpersonal relationships, Social Role (difficulties in the workplace, school or home duties)

SECONDARY OUTCOMES:
Changes in healthy eating index scores | 3 months
  Healthy eating index
General self-efficacy scale | 3 months
  Measures optimistic self-beliefs to cope with a variety of difficult demands in life.
Quick Inventory of Depressive Symptomology | 3 months
  Measures depression symptoms
Hospital Anxiety and Depression Scale | 3 months
  Measures anxiety and depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Davison, PhD, Principal Investigator — Kwantlen Polytechnic University
Locations (1):
- Innovation Boulevard, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No